CLINICAL TRIAL: NCT02204839
Title: The Metabolic and Glycaemic Effects of a Combined Basal-Bolus Insulin Reduction And Carbohydrate Feeding Strategy For Evening Exercise in Type 1 Diabetes Mellitus
Brief Title: Combined Basal-bolus Insulin and Post-exercise Carbohydrate Feeding Strategy in T1DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: West-Walker3
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM, Exercise, Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Basal dose reduction (Experimental): Total daily basal (Glargine, Lantus, Sanofi-Aventis, or Detemir, Levemir, Novo Nordisk) reduction of 20% versus normal basal dose.
  Interventions: Drug: Basal insulin dose

INTERVENTIONS:
Drug: Basal insulin dose
  Other Names: (Glargine, Lantus, Sanofi-Aventis, or Detemir, Levemir, Novo Nordisk)

SUMMARY:
The investigators hypothesise that reducing basal insulin dose (Glargine, Lantus, Sanofi-Aventis, or Detemir, Levemir, Novo Nordisk), whilst employing current carbohydrate feeding and rapid-acting insulin dose recommendations will protect patients with type 1 diabetes from early- and late-onset hypoglycaemia following evening time exercise.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-50 years old (male or female).
* Free from any diabetes related complications (apart from mild background diabetic retinopathy).
* HbA1c <8.5%.
* Not taking any prescribed medication other than insulin, and treated with a stable insulin regimen composed of a combination of slow/long acting insulin (glargine or detemir) and fast-acting insulin analogues (lispro or aspart), for a minimum of 6 months before the start of the study.
* Demonstrate normal cardiac function in response to exercise.

Exclusion Criteria:

* Aged younger than 18, or older than 50 years.
* Suffering from, or diagnosed with a diabetes related complication (apart from mild background diabetic retinopathy).
* HbA1c >8.5%.
* Currently taking prescribed medication, and not currently treated with a stable basal bolus regimen composed of a combination glargine or determir, and lispro or aspart for at least 6 months before the start of the study.
* Failure to demonstrate normal cardiopulmonary responses during exercise, or have a medical condition which could prevent completion of exercise or be exacerbated because of.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
24 hour blood glucose area under the curve | 24 hours
  24 hour blood glucose area under the curve

SECONDARY OUTCOMES:
Ketonaemia | 60 minutes before and 24 hours post-exercise
  Blood beta-hydroxybutyrate concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J West, PhD, Principal Investigator — Northumbria University
Locations (1):
- Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Campbell MD, West DJ, O'Mahoney LL, Pearson S, Kietsiriroje N, Holmes M, Ajjan RA. The relative contribution of diurnal and nocturnal glucose exposures to HbA1c in type 1 diabetes males: a pooled analysis. J Diabetes Metab Disord. 2022 Mar 31;21(1):573-581. doi: 10.1007/s40200-022-01015-1. eCollection 2022 Jun. PMID 35673512
- [Derived] Campbell MD, Walker M, Bracken RM, Turner D, Stevenson EJ, Gonzalez JT, Shaw JA, West DJ. Insulin therapy and dietary adjustments to normalize glycemia and prevent nocturnal hypoglycemia after evening exercise in type 1 diabetes: a randomized controlled trial. BMJ Open Diabetes Res Care. 2015 May 12;3(1):e000085. doi: 10.1136/bmjdrc-2015-000085. eCollection 2015. PMID 26019878